CLINICAL TRIAL: NCT00375323
Title: Effects of Recombinant Factor VIIa (NovoSeven) on Restoring Coagulation Activation in Patients With Hemophilia A and Antibodies to Factor VIII
Brief Title: Recombinant Factor VIIa (NovoSeven) on Restoring Coagulation Activation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: NovoSeven 1
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Hemophilia A
Keywords: factor VIII inhibitor
MeSH Terms: conditions — Hemophilia A | interventions — recombinant FVIIa

INTERVENTIONS:
Drug: NovoSeven

SUMMARY:
The purpose of the study is to compare the effects of recombinant factor VIIa (NovoSeven) on restoring coagulation activation between patients with hemophilia A and antibodies to factor VIII and normal subjects (controls) by use of an in vivo method.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hemophilia A and current antibodies to factor VIII -

Exclusion Criteria:

* Life-threatening hemorrhage
* Severe liver failure
* Any other severe co-morbidity (including diabetes mellitus, renal failure, cancer, septicemia, disseminated intravascular coagulation, crush injury)
* Exposure to other haemostatic drugs during the previous 7 days
* Hypersensitivity to hamster, mouse or bovine proteins
* Known or suspected allergy to NovoSeven or any of its components

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Eichinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria